CLINICAL TRIAL: NCT01067365
Title: An Open-Label, Multiple Center Study to Evaluate the Safety and Efficacy of Androxal™ Treatment in Men With Secondary Hypogonadism Who Completed ZA-003
Brief Title: Study to Evaluate the Safety and Efficacy of Androxal Treatment in Men With Secondary Hypogonadism
Acronym: ZA-003Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA-003 Extension Study
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Secondary Hypogonadism
Keywords: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12.5 mg Androxal (Experimental): 12.5 mg Androxal daily
  Interventions: Drug: Androxal
- 25 mg Androxal (Experimental): 25 mg Androxal daily
  Interventions: Drug: Androxal

INTERVENTIONS:
Drug: Androxal — 12.5 mg once daily
  Other Names: Enclomiphene citrate
  Arms: 12.5 mg Androxal
Drug: Androxal — 25 mg once daily
  Other Names: Enclomiphene citrate
  Arms: 25 mg Androxal

SUMMARY:
Subjects who completed ZA-003 were eligible to receive an additional year of treatment in this extension study.

DETAILED DESCRIPTION:
The objectives of this study were to evaluate the safety and efficacy of Androxal® administered orally once daily for one year in men with secondary hypogonadism and who had completed ZA-003.

ELIGIBILITY:
Inclusion Criteria:

* Total serum testosterone concentrations < 300 ng/dL at baseline

Exclusion Criteria:

* Presence or history of prostate cancer
* Elevated PSA > 3.5 ng/mL

Additional inclusion and exclusion criteria may apply.

Ages: 18 Years to 68 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of Androxal™ administered in men with secondary hypogonadism | One year

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (18):
- United States (18):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Medial Affiliated Research Center, Inc., Huntsville, Alabama
  - Northern California Research Corp, Carmichael, California
  - Prime-Care Clinical Research, Mission Viejo, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Commonweatlh Biomedical Research, Madisonville, Kentucky
  - The Center for Sexual Medicine at Sheppard Pratt, Baltimore, Maryland
  - Office of Keith Pierce, MD, Livonia, Michigan
  - Office of Michael Mall, MD, Las Vegas, Nevada
  - Office of Stephen Miller, MD, Las Vegas, Nevada
  - Advanced Biomedical Research, Inc., Hackensack, New Jersey
  - Office of Gary S. Karlin, MD, Lawrenceville, New Jersey
  - Medical Research Associates of Nashville, Nashville, Tennessee
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Salt Lake Research, Salt Lake City, Utah